CLINICAL TRIAL: NCT06664151
Title: A Phase 0 Window of Opportunity Trial of Intratumoral Seasonal Influenza Immunization in Cutaneous Squamous Cell Carcinoma (CSCC) Patients Awaiting Curative Excision
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Karam Khaddour, Principle Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-491
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Skin Cancer; Cutaneous Squamous Cell Carcinoma (CSCC); Cutaneous Squamous Cell Cancer
Keywords: Skin Cancer; Cutaneous Squamous Cell Carcinoma; Cutaneous Squamous Cell Cancer
MeSH Terms: conditions — Skin Neoplasms | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Fluzone Vaccine in Cutaneous Squamous Cell Carcinoma (Experimental): Enrolled participants will complete:
  * Baseline visit
  * Days 1 and 8: Flu shot injection once
  * Day 15: Standard-of-care Mohs excision surgery and tissue collection.
  * Day 21 follow up visit with suture removal.
  * Day 38 follow up visit
  Interventions: Biological: Fluzone Trivalent

INTERVENTIONS:
Biological: Fluzone Trivalent — Inactivated influenza vaccine, 0.5mL single-dose, pre-filled syringe, via intratumoral (into a tumor) injection per protocol.
  Other Names: Influenza Vaccine; Flu shot

SUMMARY:
This study is investigating the effects on immune cells of injecting the influenza vaccine (also known as "flu shot") into cutaneous squamous cell carcinoma (CSCC) tumors prior to having standard-of-care Mohs excision surgery. The study will help understand if the addition of the influenza vaccine could improve the immune system response against the cancer.

The names of the study drug involved in this study is:

-Fluzone Influenza vaccine (flu shot)

DETAILED DESCRIPTION:
This Phase 0, window-of-opportunity study is investigating the effects on immune cells of injecting the influenza vaccine (also known as "flu shot") into cutaneous squamous cell carcinoma (CSCC) tumors prior to having standard-of-care Mohs excision surgery. This study will help understand if the addition of the influenza vaccine can improve the immune system response against the cancer.

The research study procedures include screening for eligibility, in-clinic visits, blood tests, and measurements and photographs of tumors.

It is expected that 25 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of cutaneous squamous cell carcinoma that has been biopsied and confirmed histologically. Mixed histology (such as basosquamous carcinoma, sarcomatous carcinoma) is allowed.
* Participants must have a skin tumor that measures 10 - 39 mm (not less than 10 mm and not more than 39 mm) in longest dimension by clinical exam. (Participants may have more than one untreated CSCC at the time of enrollment, but only one CSCC may be treated with the study agent.)
* Participants must be candidates for treatment (excision) by Mohs micrographic surgery.
* Age ≥18 years. Because CSCC is exceptionally rare in patients <18 years of age, children are excluded from this study.
* ECOG performance status ≤3 (Karnofsky ≥40%, see Appendix A).
* Ability to understand and the willingness to sign a written informed consent document.
* For participants with a past medical history of Human immunodeficiency virus (HIV), they must be on effective anti-retroviral therapy with undetectable viral load measured within the 6 months prior to enrollment.
* For participants with a past medical history of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* For participants with a past medical history of hepatitis C virus (HCV) infection, they must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.

Exclusion Criteria:

* CSCC with the following high-risk features including peri-neural invasion of >0.1 mm caliber, and invasion of tissue beyond the subcutaneous fat, and a diameter > 3.9 cm.
* Evidence of in-transit/satellite, nodal, or distant metastases from CSCC, in the present or in the past medical history, including evidence from physical exam of primary site and draining lymph node basin.
* History of solid organ transplant or allogeneic bone marrow transplant.
* History of allergic reactions attributed to the seasonal flu vaccine.
* History of Guillain-Barré syndrome.
* Participants with any uncontrolled intercurrent illness, including uncontrolled cardiac disease (New York Heart Association Class III or IV heart failure, myocardial infarction in the 6 months prior to enrollment, unstable angina).
* Participants who are receiving any other investigational agents for treatment of cancer.
* Participants with a past medical history of another malignancy whose natural history or treatment is likely to interfere with the safety or efficacy assessment of the investigational regimen, according to the treating investigator.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of intratumoral flu vaccine administration. Patients who do not agree to comply with these precautions are ineligible.
* Pregnant or nursing (breast-feeding) women are excluded from this study because there is an unknown but potential risk to multiple injections of flu vaccine in pregnant or nursing women.
* Note: Previous treatment with flu vaccination is not an exclusion criterion. Routine intramuscular seasonal influenza vaccination is not required nor prohibited.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Mean Percent Change of CD8+ T-cells Density | Up to 15 Days
  CD8+ T-cell infiltration density (as measured by cells/mm2) on tumors is collected at the time of Mohs micrographic surgery compared to baseline (time of diagnostic biopsy).

SECONDARY OUTCOMES:
Change in Tumor Diameter | Up to 15 Days
  Evaluate the change in tumor diameter based on day 1 screening and the biopsy from the time of diagnosis.
Adverse Events | Up to 38 days
  Adverse events rate is defined as the percentage of participants who have experienced adverse events based on CTCAE 5.0
Mean Percent Change of Tumor Microenvironment Markers Compared Before and After Intratumoral Influenza Vaccination | Up to 15 Days
  Evaluation of the differences of effect on the mean percent change of tumor microenvironment markers before and after the administration of intratumoral influenza vaccine in CSCC lesions

CONTACTS AND LOCATIONS:
Overall Officials: Karam Khaddour, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu